CLINICAL TRIAL: NCT00507377
Title: Frequency, Predictors, Intraoperative Assessment and Outcome of Foreshortened Esophagus and Its Surgical Therapy in Patients Treated for Gastro-Esophageal Reflux Disease (GERD)
Brief Title: Foreshortened Esophagus and Its Surgical Therapy
Acronym: GERDSurgery
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: The European Society of Esophagology (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Other Study IDs: 61657
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Gastroesophageal Reflux Disease; Hiatal Hernia
Keywords: Esophageal Benign Disease; Gastroesophageal Reflux Disease; Hiatal Hernia; Antireflux Surgery; Short Esophagus
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background The existence, diagnosis and treatment of short esophagus is one of the controversies of the past which has recently re-emerged The missed diagnosis of short esophagus and the consequent inadequacy of treatment is one of the major causes of failure of antireflux surgery.

The daily clinical practice of surgeons dedicated to therapy of esophageal diseases could take advantage of the definition of frequency, preoperative predictors, intraoperative management and post operative outcomes of cases of foreshortened esophagus, in order to offer the patient affected by GERD the elements necessary for a conscious choice of therapy and to plan the best performance of the surgical procedure.

Aims of the Study To define the percentage of cases among the total of antireflux procedures performed, in which, after standard isolation of the ge junction and eventual dissection of the mediastinal esophagus at least two centimetres of esophagus can not be replaced without any applied tension below the apex of the diaphragmatic hiatus.

To define the percentage of surgical procedures aimed to treat electively a condition of non reducible G-E junction and foreshortened esophagus, among a multicentric formed case series of patients submitted to antireflux surgery.

To define the preoperative clinical and instrumental predictors for a surgical procedure aimed to treat foreshortened esophagus.

To record the intra-operative, postoperative, 6 month and 12 month outcome of procedures adopted for the surgical treatment of GERD.

Materials and Methods The study will comprise patients in which surgical therapy for GERD is indicated according to the international guidelines and the Centres policy .

Patients will be submitted to the antireflux procedure chosen by the surgeon according to the internationally recognized scientific surgical principles and the personal judgement.

The preoperative study and the postoperative follow up adopted in the present study are accepted by the Centres as they correspond to the international guidelines and the Centres' current practice criteria for the surgical treatment of GERD.

DETAILED DESCRIPTION:
INTRODUCTION The existence, diagnosis and treatment of short esophagus is one of the controversies of the past within esophageal surgery which has recently re-emerged. This entity was described in detail by radiologists in the 60's. Many surgeons confirmed its existence in the operating room, describing the clinical, anatomical and surgical patterns along with the modalities of surgical treatment of shortened esophagus following progressive fibrosis and retraction of the esophageal wall consequent to severe long standing gastro-esophageal reflux disease (GERD). Contrarily other surgeons denied its existence claiming that the gastro-oesophageal junction can be reduced into the abdomen without tension in virtually all patients and that the esophagus is, in fact, not shortened. In the case series of open antireflux surgery, the percentage of dedicated procedures aimed to treat the condition of non-reducibility of the gastro-esophageal junction (GEJ) below the diaphragm is highly variable.

In the present era of minimally invasive antireflux surgery, short esophagus again seems to originate controversy and open debate. Many thousands of laparoscopic standard antireflux operations have been performed in the world and numerous articles report satisfactory short and medium-term functional results in over 90% of cases, although in these experiences the need for a tailored approach has not emerged. However, in the last two or three years, many reports on the diagnosis and laparoscopic management of shortened esophagus in GERD surgery have been published.

The controversy is based on four facts.

1. If the indications for surgical therapy of GERD are restricted to severe, long standing cardial incontinence and to the complications associated with a hiatus hernia, then the number of patients with panmural esophagitis and esophageal shortening will be higher in percentage than if the indications are open also to refluxers otherwise treatable with intermittent low dosage medical therapy
2. The clinical-instrumental predictors of esophageal elastic or fibrotic shortening are not defined and current studies adopt different evaluation criteria
3. The perception of "excessive tension" of the fundoplication at the operating table is highly subjective.
4. During the process of progressive shortening of the esophagus, the portion of the fundus attracted above the diaphragm may take the appearance of a funnel hardly distinguishable from a thickened oesophagus. Therefore the gastric fundus may be erroneously wrapped around the herniated stomach.

Preoperative assessment of the length of the esophagus in order to decide which surgical technique to adopt is controversial. Yau et all. demonstrated that there is an association between esophageal shortening measured by standard manometry and postoperative para-esophageal herniation, but this increased risk is small. Predictors of the need for esophageal lengthening procedure are para-esophageal hernia, Barrett's esophagus and failed antireflux surgery. However no preoperative assessment can give information on the degree of elasticity or fibrosis of the esophagus.

Through laparoscopic surgery, by cranially distending the diaphragmatic hiatus the pneumoperitoneum may by artefact increase the length of the intra-abdominal esophagus, and the impossibility to manually palpate and feel the tension applied to the esophagus to bring the GEJ below the diaphragm may make it difficult to recognize a condition of shortened esophagus, more so if the experience of the surgeon is not adequate.

On the basis of a radiological classification used since the sixties, later validated with a radiological-manometric study it was demonstrated that the progressive orad migration of the GEJ is associated with an increasing severity of cardial incontinence and gastro-esophageal reflux.

Recent studies have shown that the permanent orad displacement of the GEJ across or above the diaphragm is not infrequent in patients affected by various grades of GERD and that it is present in 50% of patients undergoing antireflux surgery for severe, not otherwise manageable GERD. Up to 25% of patients may require a procedure of lengthening of the esophagus in order to place the fundoplication below the diaphragm without tension.

The missed diagnosis of short esophagus and the consequent inadequacy of treatment is one of the major causes of failure of antireflux surgery.

As the number of antireflux operations, mainly laparoscopic, performed per year has remarkably increased, the issue of the so-called short esophagus is today one of the major points in the management of antireflux surgery, which deserves reappraisal and definitive clarification.

The daily clinical practice of surgeons dedicated to therapy of esophageal diseases could take advantage of the definition of frequency, preoperative predictors, intraoperative management and post operative outcomes of cases of foreshortened esophagus in order to offer the patient affected by GERD, the elements necessary for a conscious choice of therapy, whether medical or surgical and to plan the best performance of the surgical procedure.

AIMS OF THE STUDY Principal aim

1. To define the percentage of cases among the total of antireflux procedures performed, in which, after standard isolation of the ge junction and eventual dissection of the mediastinal esophagus at least two centimetres of esophagus can not be replaced without any applied tension below the apex of the diaphragmatic hiatus.

   Secondary aims
2. To define the percentage of surgical procedures aimed to treat electively a condition of non reducible, foreshortened esophagus, among a multicentric formed case series of patients submitted to antireflux surgery;
3. To define the preoperative clinical and instrumental predictors for a surgical procedure aimed to treat foreshortened esophagus;
4. To record the intra-operative, postoperative, 6 month and 12 month outcome of procedures adopted for the surgical treatment of GERD;

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years, undergoing surgery for the treatment of GERD, of massive incarcerated hiatus hernia ± GERD, in which a laparotomic, laparoscopic or thoracotomic approach is preoperatively indicated.

Exclusion Criteria:

* association of GERD with epiphrenic esophageal diverticulum, collagen diseases, undetermined esophageal motility disorders;
* redo antireflux surgery, previous surgery on the thoracic and abdominal esophagus and stomach, on the diaphragm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GERD patients > 18 years
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli, MD, Study Chair — University of Bologna
Locations (8):
- Italy (8):
  - Dept. of "Surgery, Intensive Care and Organs Transplantation", Bologna
  - Department of General and Minimally Invasive Surgery -- Esophago-gastric Surgery Unit, Istituto Clinico Humanitas, Rozzano, University of Milan, Milan
  - First Division of General and Gastrointestinal Surgery, Second University of Naples, Naples
  - Unit of Gastrointestinal Surgery, School of Medicine, II University of Naples, Naples
  - VIII Division of General Surgery and Gastroenterologic Physiopathology, II University of Naples, Naples
  - Department of Medical and Surgical Sciences Clinica Chirurgica 3, University of Padova, Padua
  - General Surgery IV, Regional Referral Center for Esophageal Pathology, Department of Medical and Surgical Gastroenterology, AOU Pisana, Pisa, Pisa
  - Department of Surgery, Minimally Invasive Surgery Center, University of Turin, Turin